CLINICAL TRIAL: NCT00469248
Title: Intra-Aortic Balloon Counterpulsation in Patients With Acute Myocardial Infarction Complicated by Cardiogenic Shock - The Prospective, Randomised IABP SHOCK Trial for Attenuation of Multi-Organ Dysfunction Syndrome
Brief Title: Aortic Balloon Counterpulastion in Myocardial Infarction Related Shock
Acronym: IABPSHOCK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MLU-IABPSHOCK
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Last update posted 2007-05-04 (Estimated); Status verified 2007-04

CONDITIONS: Myocardial Infarction; Cardiogenic Shock
Keywords: Myocardial infarction; Cardiogenic shock; Systemic inflammatory response syndrome; Percutaneous coronary intervention; aortic balloon counterpulsation
MeSH Terms: conditions — Myocardial Infarction; Shock, Cardiogenic; Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Intra-aortic balloon pump counterpulsation

SUMMARY:
The role of intra aortic balloon counterpulsation in patients experiencing acute myocardial infarction with shock is not established. We hypothesised that use of such a device would lead to improved outcomes in these patients.

DETAILED DESCRIPTION:
Patients undergoing percutaneous coronary intervention (PCI) for acute myocardial infarction (AMI) with cardiogenic shock (CS) are often treated with Intra-aortic balloon pump counterpulsation (IABP) although the evidence to support this is limited. We conducted a prospective, randomised clinical trial, of IABP as an addition to PCI centred therapy, in patients with AMI complicated by CS.

45 patients with AMI and CS undergoing PCI were randomised to care with or without IABP. Over 4 days, APACHE II scores, haemodynamic parameters, inflammatory markers and BNP levels were collected to assess the impact of IABP treatment on CS triggered multi organ dysfunction syndrome (MODS).

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction
* Cardiogenic shock

Exclusion Criteria:

* Absent peripheral pulses
* Mechanical complications of myocardial infarction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2003-03; Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
APACHE II SCORE | 4 days

SECONDARY OUTCOMES:
Haemodynamic state | 4 days
BNP levels | 4 days
Inflammatory activation | 4 days
Mortality | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Buerke, MD, Study Chair — Martin Luther University; Roland Prondzinsky, MD, Principal Investigator — Martin Luther University
Locations (1):
- Department of Medicine III, Klinikum Krollwitz, Martin Luther University, Halle, Saxony-Anhalt, Germany

REFERENCES:
- [Derived] Prondzinsky R, Unverzagt S, Lemm H, Wegener N, Heinroth K, Buerke U, Fiedler M, Thiery J, Haerting J, Werdan K, Buerke M. Acute myocardial infarction and cardiogenic shock: prognostic impact of cytokines: INF-gamma, TNF-alpha, MIP-1beta, G-CSF, and MCP-1beta. Med Klin Intensivmed Notfmed. 2012 Sep;107(6):476-84. doi: 10.1007/s00063-012-0117-y. Epub 2012 Jul 20. PMID 22810435
- [Derived] Prondzinsky R, Unverzagt S, Russ M, Lemm H, Swyter M, Wegener N, Buerke U, Raaz U, Ebelt H, Schlitt A, Heinroth K, Haerting J, Werdan K, Buerke M. Hemodynamic effects of intra-aortic balloon counterpulsation in patients with acute myocardial infarction complicated by cardiogenic shock: the prospective, randomized IABP shock trial. Shock. 2012 Apr;37(4):378-84. doi: 10.1097/SHK.0b013e31824a67af. PMID 22266974
- [Derived] Prondzinsky R, Unverzagt S, Lemm H, Wegener NA, Schlitt A, Heinroth KM, Dietz S, Buerke U, Kellner P, Loppnow H, Fiedler MG, Thiery J, Werdan K, Buerke M. Interleukin-6, -7, -8 and -10 predict outcome in acute myocardial infarction complicated by cardiogenic shock. Clin Res Cardiol. 2012 May;101(5):375-84. doi: 10.1007/s00392-011-0403-3. Epub 2012 Jan 3. PMID 22212516
- [Derived] Prondzinsky R, Lemm H, Swyter M, Wegener N, Unverzagt S, Carter JM, Russ M, Schlitt A, Buerke U, Christoph A, Schmidt H, Winkler M, Thiery J, Werdan K, Buerke M. Intra-aortic balloon counterpulsation in patients with acute myocardial infarction complicated by cardiogenic shock: the prospective, randomized IABP SHOCK Trial for attenuation of multiorgan dysfunction syndrome. Crit Care Med. 2010 Jan;38(1):152-60. doi: 10.1097/CCM.0b013e3181b78671. PMID 19770739